CLINICAL TRIAL: NCT00004488
Title: Phase II Randomized Study of Alendronate Sodium for Osteopenia in Patients With Gaucher's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 199/14269; CHMC-C-FDR001537; CHMC-C-498
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-03

CONDITIONS: Gaucher's Disease; Osteopenia
Keywords: Gaucher's disease; inborn errors of metabolism; rare disease; sphingolipidoses
MeSH Terms: conditions — Gaucher Disease; Bone Diseases, Metabolic; Metabolism, Inborn Errors; Rare Diseases; Sphingolipidoses | interventions — Alendronate; Calcium Carbonate; Cholecalciferol

INTERVENTIONS:
Drug: alendronate sodium
Drug: calcium carbonate
Drug: cholecalciferol

SUMMARY:
OBJECTIVES:

I. Determine the efficacy of alendronate sodium in treating osteopenia (generalized bone density and focal bone lesions) in patients with Gaucher's disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, double blind, placebo controlled study.

All patients receive oral calcium carbonate and cholecalciferol daily. Patients are randomized to receive oral alendronate sodium or placebo daily for 24 months.

Patients are followed every 6 months for 2 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Diagnosis of type 1 Gaucher's disease enzymatically proven to have acid beta glucosidase deficiency

Must have been on stable dose (8-60 U/kg/every 2 weeks) of alglucerase enzyme therapy (Cerezyme or Ceredase) for at least 24 months

Lumbar spine bone density below the mean for age, sex, and race

--Prior/Concurrent Therapy--

At least 6 months since prior medications that directly affect skeletal metabolism including, but not limited to, bisphosphonates, calcitonin, parathyroid hormone, or estrogen

--Patient Characteristics--

Renal: No chronic renal failure; No recurrent renal stones

Esophageal: No history of dysphagia; No frequent heartburn; No esophagitis requiring treatment

Other: No untreated hyperthyroidism or hypothyroidism; No concurrent hyperparathyroidism; No concurrent malignancy; No history of alcohol or drug abuse; Not pregnant; Negative pregnancy test; Fertile patients must use effective contraception

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Estimated)
Dates: Start 1998-10; Study Completion 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Wenstrup, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (2):
  - Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio
  - Wright State University School of Medicine, Dayton, Ohio
- Shaare Zedek Medical Center, Jerusalem, Israel